CLINICAL TRIAL: NCT04186520
Title: Phase I/II Study of Tandem, Bispecific Anti-CD19 Anti-CD20 CAR-T Cells for Patients With Relapsed and/or Refractory B Cell Malignancies
Brief Title: CAR-20/19-T Cells in Patients With Relapsed Refractory B Cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nirav Shah, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037171
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Non Hodgkin Lymphoma (NHL); Mantle Cell Lymphoma (MCL); Chronic Lymphocytic Leukemia (CLL); Follicular Lymphoma; Marginal Zone Lymphoma; Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Central Nervous System Lymphoma
Keywords: CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy; B-cell Malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 8/12 Day Production of CAR-T for NHL (Experimental): Phase 1: Determine safety of 2.5x10^6 cells/kg IL-7/IL-15 expanded CAR-20/19-T cells in patients with relapsed, refractory B-cell NHL. Patients will be enrolled in 3+3 fashion.
  Phase 1b: Six to nine patient expansion cohorts at eight or 12-day manufacturing. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12 in each group.
  Interventions: Biological: 8/12-Day Production of Car-T Cells
- 8/12 Day Production of CAR-T for CLL (Experimental): Phase 1: Determine safety of 2.5x10^6 cells/kg IL-7/IL-15 expanded CAR-20/19-T cells in patients with CLL. Patients will be enrolled in 3+3 fashion.
  Phase 1b: The enrollment will cap at 24 subjects.
  Interventions: Biological: 8/12-Day Production of Car-T Cells
- 8/12 Flexible Manufacturing with Mandated Cryopreservation (Experimental): 8/12 flexible manufacturing with mandated cryopreservation prior to infusion of LV20.19 CAR T-cells. The enrollment will cap at 24 subjects.
  Interventions: Biological: 8/12-Day Production of Cryopreserved Car-T Cells
- 12-Day Production of Car-T Cells for NHL (Experimental): Phase 1: Determine safety of 2.5x10^6 cells/kg IL-7/IL-15 expanded CAR-20/19-T cells in patients with relapsed, refractory B-cell NHL. Patients will be enrolled in 3+3 fashion.
  Phase 1b: Six to nine patient expansion cohorts at 12-day manufacturing. If six patients are enrolled in Phase 1 then only six additional patients will be added. If three patients are enrolled in Phase 1 then nine additional patients will be treated for a total of 12 in each group.
  Interventions: Biological: 12-Day Production of Car-T Cells
- 8/12 Day Production of CAR-T for Relapsed/Refractory Primary or Secondary CNS Lymphoma (Experimental): Phase 1: Determine safety of 2.5x106 cells/kg IL-7/IL-15 expanded CAR-20/19-T cells in patients with primary/secondary central nervous system (CNS) lymphoma.
  Phase 1b: Safety and efficacy will be evaluated in this study that will enroll 12 to 24 patients.
  Interventions: Biological: 8/12-Day Production of Car-T Cells
- Phase 2 - Efficacy of CAR-20/19-T cells in MCL (Experimental): Single-stage Phase II design with three-month CR as the target endpoint.
  Interventions: Biological: 8/12-Day Production of Car-T Cells

INTERVENTIONS:
Biological: 8/12-Day Production of Car-T Cells — A fixed dose of 2.5 x 10^6 CAR-20/19-T cells/kg expanded with IL-7/IL-15.
  Arms: 8/12 Day Production of CAR-T for CLL; 8/12 Day Production of CAR-T for NHL; 8/12 Day Production of CAR-T for Relapsed/Refractory Primary or Secondary CNS Lymphoma; Phase 2 - Efficacy of CAR-20/19-T cells in MCL
Biological: 8/12-Day Production of Cryopreserved Car-T Cells — A fixed cryopreserved dose of 2.5 x 10^6 CAR-20/19-T cells/kg expanded with IL-7/IL-15.
  Arms: 8/12 Flexible Manufacturing with Mandated Cryopreservation
Biological: 12-Day Production of Car-T Cells — A fixed dose of 2.5 x 10^6 CAR-20/19-T cells/kg expanded with IL-7/IL-15.
  Arms: 12-Day Production of Car-T Cells for NHL

SUMMARY:
This is a Phase I/II, interventional, single-arm, open-label, treatment study designed to evaluate the safety and efficacy of Interleukin-7 and Interleukin-15 (IL-7/IL-15) manufactured chimeric antigen receptor (CAR)-20/19-T cells as well as the feasibility of a flexible manufacturing schema in adult patients with B cell malignancies that have failed prior therapies.

DETAILED DESCRIPTION:
This is a Phase 1/Phase 2 study. The objectives are as follows:

1. Phase 1: Determine the safety of a fixed dose of 2.5x10^6 CAR-20/19-T cells/kg expanded with IL-7/IL-15 in relapsed refractory B-cell NHL with flexible 8/12-day manufacturing and a fixed 12-day manufacturing process along with an evaluation in chronic lymphocytic leukemia (CLL) and central nervous system (CNS) lymphoma.
2. Phase 1b: Four arms:

   Arm A: 8/12 flexible manufacturing arm. Determine safety, efficacy, and feasibility of flexible manufacturing.

   Arm B: Fixed 12-day manufacturing arm. Determine safety and efficacy of fixed CAR manufacturing.

   Arm C: 8/12 flexible manufacturing with mandated cryopreservation prior to infusion of LV20.19 CAR T-cells. Determine the impact of cryopreservation on safety or efficacy of LV20.19 CAR T-cells.

   Arm D: 8/12 flexible manufacturing expansion cohort in CLL. Determine safety and efficacy in CLL.

   Arm E: 8/12 flexible manufacturing cohort in central nervous system (CNS) lymphoma.
3. Phase 2

   1. Determine the 3-month CR rate of CAR-20/19-T cells in MCL
   2. Determine the feasibility of a flexible manufacturing process of CAR-20/19-T cells from patient apheresis products using the CliniMACS Prodigy Cell processing device

ELIGIBILITY:
GENERAL INCLUSION CRITERIA FOR ALL PATIENTS

1. Patients must be aged ≥18 years and ≤80 years with relapsed or refractory B-cell non-Hodgkin Lymphoma.
2. Absolute cluster of differentiation 3 (CD3) count ≥50 mm^3.
3. Magnetic resonance imaging (MRI) brain and lumbar puncture with cerebrospinal fluid (CSF) analysis by cytology and flow cytometry without evidence of central nervous system (CNS) involvement ONLY in patients with history of CNS involvement or clinical suspicion at the time of enrollment EXCEPT Arm E subjects.
4. Measurable disease must be documented within four weeks of the time of consent defined as nodal lesions greater than 15 mm in the long axis or extranodal lesions >10 mm in long and short axis OR bone marrow involvement that is biopsy proven for B-cell NHL (see separate criteria for CLL and primary/secondary CNS lymphoma).
5. Karnofsky performance score ≥70.
6. Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <5 x upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <5 x ULN, or considered not clinically significant as per the clinical PIs discretion (e.g. Gilbert's or indirect hyperbilirubinemia) or felt to be due to underlying disease.
7. ANC≥1000 with no G-CSF within 72 hours or pegylated G-CSF within 14 days.
8. Platelets≥50,000 with no transfusion within 72 hours.
9. Adequate renal function, defined as creatinine clearance >60 ml/min AND serum Cr≤1.5 mg/dL.

   a. No IV hydration within 24 hours of eligibility. b. No dialysis dependent renal failure within three months of planned CAR infusion.
10. Able to provide written informed consent.
11. Agree to practice birth control during the study.
12. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥45% (by cardiac echocardiogram (ECHO) or multigated acquisition scan (MUGA)) and adequate pulmonary function as indicated by room air oxygen saturation of ≥92%.
13. Expected survival >12 weeks.
14. Negative urine or serum pregnancy test in females of child bearing potential at study entry.
15. Meet criteria regarding fertility and contraception.
16. No contraindication to central line access.
17. Patient has demonstrated compliance to other therapies.

Phase 1: 3+3 COHORT ELEGIBILITY CRITERIA

1. Diagnosis of B-cell NHL including Follicular Lymphoma, Marginal Zone Lymphoma (splenic, nodal, extranodal), Mantle Cell Lymphoma, and DLBCL with associated subtypes (aggressive B-cell lymphoma, high grade B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, Epstein-Barr virus-positive (EBV+) diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).
2. Patients must have active, measurable disease as defined and meet one of the following criteria.

   1. Must have received Rituximab or another cluster of differentiation 20 (CD20) antibody and at minimum two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant.
   2. Relapse post-autologous transplant
   3. Relapse post-allogeneic transplant
   4. Patients not previously treated with CAR-T cell therapy

PHASE 1b and 2 COHORT ELEGIBILITY CRITERIA

ARM A: Six to nine patient expansion with 8-day manufacturing (Phase 1b)

1. Diagnosis of B-cell NHL including Follicular Lymphoma, Marginal Zone Lymphoma (splenic, nodal, extranodal), and DLBCL with associated subtypes (aggressive B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, EBV+ diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).
2. Patients must have active, measurable disease as defined and meet one of the following criteria:

   1. Must have received Rituximab or another cluster of differentiation 20 (CD20) antibody and at minimum two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant.
   2. Relapse post-autologous transplant.
   3. Relapse post-allogeneic transplant.
   4. Relapse post-anti-cluster of differentiation 19 (CD19) CAR-T cell therapy.

   i. A maximum of two patients with prior CAR-T will be allowed in this cohort.

ARM B: Six to nine patient expansion with 12-day manufacturing (Phase 1b)

1. Diagnosis of B-cell NHL including Follicular Lymphoma, Marginal Zone Lymphoma (splenic, nodal, extranodal), and DLBCL with associated subtypes (aggressive B-cell lymphoma, high grade B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, EBV+ diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).

2. Patients must have active, measurable disease as defined and meet one of the following criteria:

1. Must have received Rituximab or another CD20 antibody and at minimum two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant.
2. Relapse post-autologous transplant.
3. Relapse post-allogeneic transplant.
4. Relapse post-anti-CD19 CAR-T cell therapy.

i. A maximum of two patients with prior CAR-T will be allowed in this cohort.

ARM C: 24 patient cryopreservation 8/12 flexible manufacturing arm

1. Diagnosis of B-cell NHL including Follicular Lymphoma, Marginal Zone Lymphoma (splenic, nodal, extranodal), and DLBCL with associated subtypes (aggressive B-cell lymphoma, high grade B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, EBV+ diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).
2. Patients must have active, measurable disease as defined and meet one of the following criteria a. Must have received Rituximab or another CD20 antibody and at minimum two different chemotherapy regimens appropriate for their disease and be ineligible to receive autologous transplant b. Relapse post-autologous transplant c. Relapse post-allogeneic transplant d. Relapse post-anti-CD19 CAR-T cell therapy i. A maximum of 2 patients with prior CAR-T will be allowed in this cohort

ARM D: Phase 1 and Phase 1b: CLL

1. Diagnosis of B-cell CLL or small lymphocytic leukemia (SLL) 2. Failed/progressed or been intolerant to two prior lines of therapy one of which MUST be either a covalent BTK inhibitor (e.g. ibrutinib, acalabrutinib, zanabrutinib, etc) or BCL2 inhibitors (e.g. venetoclax or other investigational BCL2) 3. Indication for treatment as defined as any of the following:

1. measurable lymph nodes ≥ 1.5 cm in the greatest transverse diameter and/or hepatomegaly or splenomegaly)
2. bone marrow involvement with ≥10% CLL involvement

ARM E: Phase 1 and Phase1b Relapsed/Refractory Primary or Secondary CNS Lymphoma

1. Diagnosis of diffuse large B cell lymphoma (DLBCL) with associated subtypes (aggressive B-cell lymphoma, high grade B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, EBV+ diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation) with secondary CNS lymphoma involvement OR primary CNS lymphoma.
2. For Primary CNS lymphoma, relapsed or refractory following at least one line of CNS-directed therapy.
3. Secondary CNS lymphoma relapsed or refractory following at least one line of CNS-directed therapy for treatment of CNS lymphoma.

   1. For patients with secondary central nervous system lymphoma (CNSL) with concurrent systemic lymphoma, the concurrent systemic lymphoma must have relapsed following at least 1 prior line of therapy (which must have included an anti-CD20 monoclonal antibody and an anthracycline)
4. Measurable CNS disease by either lumbar puncture (LP) with positivity in CNS by flow cytometry or morphology for lymphoma cells OR magnetic resonance imaging (MRI) with enhancing lesions ≥1 cm in size consistent with lymphoma
5. Must have had prior treatment with high dose methotrexate defined as methotrexate given intravenously at a dose ≥2500 mg/m^2 and either progression/relapse, stable disease, or intolerance to at least one cycle of treatment.

Phase II Cohort: Mantle Cell Lymphoma

1. Diagnosis of Mantle Cell Lymphoma. 2. Patients must have active, measurable disease as previously defined and have relapsed, refractory disease as defined as one of the following:

1. Relapsed disease after two lines of cytotoxic chemotherapy including administration of anti-CD20 antibody.
2. Progressive disease after ≥second line Bruton tyrosine kinase (BTK) inhibitor.
3. Relapse post-autologous transplant.
4. Relapse post-allogeneic transplant.
5. Relapse post anti-CD19 CAR-T cell therapy.

i. A maximum of four patients with history of prior anti-CD19 CAR-T will be allowed in this cohort.

EXCLUSION CRITERIA (ALL PATIENTS)

A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Positive beta- human chorionic gonadotropin (HCG) in female of childbearing potential.
2. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
3. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
4. Presence of ≥grade 3 non-hematologic toxicities as per CTCAE version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
5. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution. Minimum of 14 days or 5 half-lives of the drug (whichever is shorter) washout prior to apheresis.
6. Refusal to participate in the long-term follow-up protocol
7. Patients with active CNS involvement by malignancy on MRI or by lumbar puncture (Not applicable to Arm E cohort.)

   a. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment and a remission documented within 8 weeks of planned CAR-T cell infusion by MRI brain and CSF analysis.
8. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <100 days' post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
9. Prior allogeneic CAR T-cell therapy
10. Previous recipients of autologous CAR-T cell therapy directed at either CD19 or CD20 are excluded if they are <100 days post prior CAR-T cell treatment (does not include re-enrollment) or have >5% residual circulating CAR-T as measured by flow cytometry using a CD19 CAR detection reagent (Miltenyi Biotec)

    a. Patients with prior CAR-T treatment against CD19 or CD20 must have repeat biopsy post-CAR-T cell therapy confirming a minimum of 5% CD19 or CD20 positivity by immunohistochemistry or flow cytometry
11. Anti-CD20 antibody treatment within 4 weeks of cell infusion
12. Anti-CD19 antibody treatment within 4 weeks of cell infusion
13. Cytotoxic chemotherapy other than lymphodepletion within 14 days of CAR-T cell infusion
14. Cytotoxic chemotherapy treatment within 14 days or steroid treatment (other than replacement dose steroids) within 7 days prior to apheresis collection for CAR-T cells
15. Oral chemotherapeutic agents or antibody directed treatment within 7 days of apheresis

    a. BTK inhibitors are allowed until 1-day prior to apheresis and can re-start until 1-day prior to lymphodepletion
16. Patients post solid organ transplant who develop high grade lymphomas or leukemias
17. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin (underlying low-grade lymphoma chronic lymphocytic leukemia/follicular lymphoma (FL)/marginal zone lymphoma (MZL) is allowable in patients with transformed large cell lymphoma)

SPECIAL CRITERIA REGARDING FERTILITY AND CONTRACEPTION

Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed as part of eligibility criteria Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception during the follow-up period of the protocol.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormonal-based contraception Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events after CAR 20/19-T cell infusion | Within the first 28 days after infusion
  Incidence of adverse events using NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah NN, Colina AS, Johnson BD, Szabo A, Furqan F, Kearl T, Schneider D, Vargas-Cortes M, Schmeling JL, Dwinell MB, Palen K, Longo W, Hematti P, Zamora AE, Hari P, Bucklan D, Cunningham A, Hamadani M, Fenske TS. Phase I/II Study of Adaptive Manufactured Lentiviral Anti-CD20/Anti-CD19 Chimeric Antigen Receptor T Cells for Relapsed, Refractory Mantle Cell Lymphoma. J Clin Oncol. 2025 Jul 10;43(20):2285-2295. doi: 10.1200/JCO-24-02158. Epub 2025 Mar 31. PMID 40163793
- [Derived] Zurko JC, Xu H, Chaney K, Schneider D, Szabo A, Hari P, Johnson BD, Shah NN. Bispecific targeting of CD20 and CD19 increases polyfunctionality of chimeric antigen receptor T-cell products in B-cell malignancies. Cytotherapy. 2022 Aug;24(8):767-773. doi: 10.1016/j.jcyt.2022.03.011. Epub 2022 May 18. PMID 35597752